CLINICAL TRIAL: NCT03320213
Title: Value of CA125 and Yolk Sac Morphology in Prediction of Pregnancy Outcome in Threatened Miscarriage
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Mahmoud Sami, gynecology and obstetrics resident at ministry of health and population, Ain Shams University
Other Study IDs: 136
Record Dates: First submitted 2017-10-08; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Threatened Miscarriage in First Trimester
Keywords: CA125; Yolk sac morphology; Threatened miscarriage
MeSH Terms: conditions — Abortion, Threatened

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
evaluation of serum CA125 level and yolk sac morphology in women with threatened miscarriage is very important to predict pregnancy outcome

ELIGIBILITY:
Inclusion Criteria:

* pregnant women between 20-40 years. Pregnancy between 6-10 weeks. single intrauterine spontaneous pregnancy. vaginal bleeding or bloody vaginal discharge with or without pelvic pain for patients with threatened miscarriage.

Exclusion Criteria:

* medical disorders with pregnancy. History of recurrent miscarriage. Any maternal disease that would cause an increase in CA125 level. Local gynecological disorders e.g. fibroid. Presence of any uterine malformation. History of congenital abnormalities in previous pregnancy Presence of multiple pregnancy. Presence of anembryonic sac. Absent fetal heart pulsation.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women at age of 20- 40 years Pregnancy at 6-10 weeks women with single intrauterine spontaneous pregnancy
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of serum CA125 | 6 - 10 weeks
  Measuring serum level of CA125 by ELIZA kits.
Evaluation of yolk sac morphology | 6 - 10 weeks
  Evaluating yolk sac size and shape by transvaginal ultrasound

SECONDARY OUTCOMES:
follow up of participants | up to 20 weeks
  measuring fetal heart rate by transvaginal ultrasound.
follow up of participants | up to 20 weeks.
  measuring crown rump length by transvaginal ultrasound.